CLINICAL TRIAL: NCT02679755
Title: A STUDY OF PALBOCICLIB IN COMBINATION WITH LETROZOLE AS TREATMENT OF POST-MENOPAUSAL WOMEN WITH HORMONE RECEPTOR-POSITIVE, HER2-NEGATIVE ADVANCED BREAST CANCER FOR WHOM LETROZOLE THERAPY IS DEEMED APPROPRIATE
Brief Title: Palbociclib In Combination With Letrozole As Treatment Of Post-Menopausal Women With HR+, HER2- Advanced Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A5481037
Record Dates: First submitted 2016-01-22; First posted 2016-02-10 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Hormone receptor positive advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): Palbociclib plus Letrozole
  Interventions: Drug: Palbociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — 125 mg/d capsules orally for 3 out of 4 weeks in repeated cycles
  Other Names: IBRANCE
Drug: Letrozole — 2.5 mg/d tablets orally on a continuous regimen

SUMMARY:
A study of palbociclib in combination with letrozole as treatment of post-menopausal women with hormone receptor-positive, her2-negative advanced breast cancer for whom letrozole therapy is deemed appropriate.

DETAILED DESCRIPTION:
To provide access to palbociclib to post-menopausal patients with hormone receptor-positive [HR(+)], HER2-negative [HER2(-)] ABC who are deemed appropriate for letrozole therapy.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (>=18 years of age) with proven diagnosis of advanced carcinoma of the breast (ER(+) and/or PgR(+) and HER2(-)) who are appropriate for letrozole therapy (in the first-line advanced/metastatic disease setting).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate bone marrow, liver, and renal function.

Exclusion Criteria:

* Prior treatment with any CDK inhibitor .
* QTc >480 msec; history of QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes.
* High cardiovascular risk, including, but not limited to myocardial infarction, severe/unstable angina, severe cardiac dysrhythmias, and symptomatic pulmonary embolism in the past 6 months of enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 252 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- Australia (22):
  - Benjamin Carl Forster, North Sydney, New South Wales
  - Dr. Alexander Maxwell Menzies, North Sydney, New South Wales
  - HPS Pharmacies - North Sydney, North Sydney, New South Wales
  - Mater Hospital Sydney, North Sydney, New South Wales
  - Professor Frances Mary Boyle, North Sydney, New South Wales
  - Royal North Shore Hospital - Clinical Trials Pharmacy, St Leonards, New South Wales
  - Royal North Shore Hospital, Dept. of Medical Oncology, St Leonards, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - River City Pharmacy, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Care, Corporate Office, South Brisbane, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Flinders Medical Centre-Pharmacy Department, Bedford Park, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre Pharmacy, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital Pharmacy, St Albans, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Pharmacy Department, Murdoch, Western Australia
- India (12):
  - The Gujarat Cancer & Research Institute, M.P Shah Cancer Hospital, Ahmedabad, Gujarat
  - Manipal Hospital, Bangalore, Karnataka
  - HealthCare Global Enterprises Ltd., Bangalore, Karnataka
  - Kasturba Hospital, Manipal, Karnataka
  - Tata Memorial Centre, Tata Memorial Hospital, Mumbai, Maharashtra
  - Meditrina Institute Of Medical Sciences, Nagpur, Maharashtra
  - Shatabdi Hospital, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Center, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Dr. B.R.A Institute Rotary Cancer Hospital, All India Institue of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Apollo Speciality Hospital, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 252 participants were assigned to treatment at 20 sites in India and Australia (100 in India, 152 in Australia)
Groups:
- Palbociclib+Letrozole India Cohort; Palbociclib+Letrozole Australia Cohort: Participants received Palbociclib orally once a day at 125 mg for 21 days followed by 7 days off treatment for each 28-day cycle. Participants received Letrozole orally at 2.5 mg once daily as continuous daily dosing schedule according to product labeling and in compliance with its local prescribing information
Period: Overall Study
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort
Started | 100 | 152
Completed | 66 | 47
Not Completed | 34 | 105
Not completed — Death | 0 | 3
Not completed — Global deterioration of health status | 1 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Objective progression or relapse | 24 | 83
Not completed — Not defined | 0 | 2
Not completed — Withdrawal by participant | 6 | 3
Not completed — Adverse Event | 1 | 4
Not completed — Adverse events not related to study drug | 1 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Total
Number analyzed (Participants) | 100 | 152 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 107 | 178
  >=65 years | 29 | 45 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 152 | 252
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 100 | 12 | 112
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 130 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. All AEs reported after initiation of study drug treatment were considered as treatment emergent adverse events (TEAEs). AE severity was graded according to Common Terminology Criteria for AEs (CTCAE) version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 28 days after last dose of study treatment, an average of 14 months
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Palbociclib+Letrozole India Cohort; Palbociclib+LetrozoleTotal: Participants received Palbociclib orally once a day at 125 mg for 21 days followed by 7 days off treatment ofr each 28-day cycle. Participants received Letrozole orally at 2.5 mg once daily as continuous daily dosing schedule according to product labeling and in compliance with its local prescribing information
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+LetrozoleTotal
Number analyzed (Participants) | 100 | 152 | 252
Participants
  Participants with adverse events | 92 | 152 | 244
  Participants with serious adverse events | 18 | 45 | 63
  Participants with grade 3 or 4 adverse events | 69 | 124 | 193
  Participants with grade 5 adverse events | 3 | 7 | 10
  Participants discontinued due to adverse events | 2 | 9 | 11

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity (All Causalities)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. All AEs reported after initiation of study drug treatment were considered as TEAE. AE severity was graded according to Common Terminology Criteria for AEs (CTCAE) version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity.
Time Frame: Baseline up to 28 days after last dose of study treatment, an average of 14 months
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Palbociclib+Letrozole Total: Participants received Palbociclib orally once a day at 125 mg for 21 days followed by 7 days off treatment ofr each 28-day cycle. Participants received Letrozole orally at 2.5 mg once daily as continuous daily dosing schedule according to product labeling and in compliance with its local prescribing information
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+Letrozole Total
Number analyzed (Participants) | 100 | 152 | 252
Participants
  Grade 1 | 7 | 11 | 18
  Grade 2 | 16 | 16 | 32
  Grade 3 | 49 | 105 | 154
  Grade 4 | 17 | 13 | 30
  Grade 5 | 3 | 7 | 10

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Palbociclib-Related)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. All AEs reported after initiation of study drug treatment were considered as TEAE. AE severity was graded according to Common Terminology Criteria for AEs (CTCAE) version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Palbociclib-related TEAEs were determined by the investigator.
Time Frame: Baseline up to 28 days after last dose of study treatment, an average of 14 months
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+Letrozole Total
Number analyzed (Participants) | 100 | 152 | 252
Participants
  Participants with adverse events | 80 | 143 | 223
  Participants with serious adverse events | 8 | 12 | 20
  Participants with grade 3 or 4 adverse events | 64 | 108 | 172
  Participants with grade 5 adverse events | 0 | 1 | 1
  Participants discontinued due to adverse events | 1 | 4 | 5

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity (Palbociclib-Related)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. All AEs reported after initiation of study drug treatment were considered as TEAE. AE severity was graded according to Common Terminology Criteria for AEs (CTCAE) version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity. Palbociclib-related TEAEs were determined by the investigator.
Time Frame: Baseline up to 28 days after last dose of study treatment, an average of 14 months
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+Letrozole Total
Number analyzed (Participants) | 100 | 152 | 252
Participants
  Grade 1 | 6 | 21 | 27
  Grade 2 | 10 | 14 | 24
  Grade 3 | 49 | 93 | 142
  Grade 4 | 15 | 14 | 29
  Grade 5 | 0 | 1 | 1

5. Primary Outcome: Number of Participants With Serious Adverse Events (All Causalities and Palbociclib-Related)
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Palbociclib-related SAEs were determined by the investigator.
Time Frame: Baseline up to 28 days after last dose of study treatment, an average of 14 months
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+Letrozole Total
Number analyzed (Participants) | 100 | 152 | 252
Participants
  All-causality | 18 | 45 | 63
  Palciclib-Related | 8 | 12 | 20

6. Secondary Outcome: Percentage of Participants With Complete Response and Partial Response
Description: Tumor response assessments were evaluated as per local guidelines by investigators and were collected in the CRF. No response confirmation was applied.
Time Frame: Baseline and per routine clinical practice to time of last dose of study treatment, an average of 1 year
Population: The analysis population included participants with efficacy data contributing to the analysis
Measure: Number; unit: Percentage of evaluable participants
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+Letrozole Total
Number analyzed (Participants) | 100 | 152 | 252
Percentage of evaluable participants
  Percentage of participants with complete response | 1.0 | 1.3 | 1.2
  Percentage of participants with partial response | 28.0 | 11.8 | 18.3

7. Secondary Outcome: The Objective Response Rate (ORR)
Description: The tumor response was based on the response reported by investigator per local practice. No response confirmation was applied. ORR was defined as the percentage of participants with complete response or partial response relative to all as-treated population.
Time Frame: Baseline and per routine clinical practice to time of last dose of study treatment, an average of 1 year
Population: The analysis population included participants with efficacy data contributing to the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of evaluable participants
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort | Palbociclib+Letrozole Total
Number analyzed (Participants) | 100 | 152 | 252
Percentage of evaluable participants | 29.0 [20.4 to 38.9] | 13.2 [8.2 to 19.6] | 19.4 [14.7 to 24.9]

8. Secondary Outcome: EQ-5D Health Utility Index Score
Description: The EuroQol-5D (EQ-5D) (version 3L) consisted of 2 parts. The first part was a 5 item questionnaire designed to assess health status in terms of a single index value or utility score. It consisted of 5 descriptors of current health state (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). A respondent was asked to rate each state on a three level scale (1=no problem, 2=some problem, and 3=extreme problem) with higher levels indicating greater severity/impairment. The answers given to the 5 descriptors permit to find 243 unique health states which can be converted into a single EQ-5D index value by published algorithms. For the EQ-5D index, published weights are available that allow for the creation of a summary score ranging from -0.594 to 1, with low scores representing a higher level of dysfunction and 1 as perfect health.
Time Frame: The descriptive analysis was carried out on Day 1 of each cycle (cycle 1 to cycle 38), at end of treatment (EOT) and end of study (EOS), up to 3 years. Cycle 1 Day 1 is taken to be baseline.
Population: Patient reported outcome (PRO)-evaluable population was only consisted of the Australia cohort
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort
Number analyzed (Participants) | 0 | 146
Scores on a scale
  Cycle 1 Day 1 |  | 0.786 (0.171)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 139
  Cycle 2 Day 1 |  | 0.798 (0.187)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 132
  Cycle 3 Day 1 |  | 0.798 (0.169)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 119
  Cycle 4 Day 1 |  | 0.836 (0.172)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 113
  Cycle 5 Day 1 |  | 0.838 (0.153)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 106
  Cycle 6 Day 1 |  | 0.825 (0.185)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 105
  Cycle 7 Day 1 |  | 0.818 (0.167)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 97
  Cycle 8 Day 1 |  | 0.831 (0.169)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 94
  Cycle 9 Day 1 |  | 0.845 (0.149)
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 94
  Cycle 10 Day 1 |  | 0.840 (0.162)
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 88
  Cycle 11 Day 1 |  | 0.820 (0.193)
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 84
  Cycle 12 Day 1 |  | 0.810 (0.188)
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 79
  Cycle 13 Day 1 |  | 0.839 (0.183)
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 79
  Cycle 14 Day 1 |  | 0.842 (0.159)
  Cycle 15 Day 1: number analyzed (Participants) | 0 | 74
  Cycle 15 Day 1 |  | 0.840 (0.138)
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 16 Day 1 |  | 0.830 (0.182)
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 17 Day 1 |  | 0.837 (0.163)
  Cycle 18 Day 1: number analyzed (Participants) | 0 | 66
  Cycle 18 Day 1 |  | 0.836 (0.182)
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 62
  Cycle 19 Day 1 |  | 0.848 (0.179)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 61
  Cycle 20 Day 1 |  | 0.853 (0.143)
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 57
  Cycle 21 Day 1 |  | 0.868 (0.132)
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 53
  Cycle 22 Day 1 |  | 0.864 (0.132)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 48
  Cycle 23 Day 1 |  | 0.846 (0.170)
  Cycle 24 Day 1: number analyzed (Participants) | 0 | 42
  Cycle 24 Day 1 |  | 0.864 (0.135)
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 36
  Cycle 25 Day 1 |  | 0.861 (0.138)
  Cycle 26 Day 1: number analyzed (Participants) | 0 | 31
  Cycle 26 Day 1 |  | 0.869 (0.143)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 27
  Cycle 27 Day 1 |  | 0.884 (0.140)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 24
  Cycle 28 Day 1 |  | 0.876 (0.152)
  Cycle 29 Day 1: number analyzed (Participants) | 0 | 21
  Cycle 29 Day 1 |  | 0.852 (0.147)
  Cycle 30 Day 1: number analyzed (Participants) | 0 | 18
  Cycle 30 Day 1 |  | 0.857 (0.160)
  Cycle 31 Day 1: number analyzed (Participants) | 0 | 16
  Cycle 31 Day 1 |  | 0.784 (0.278)
  Cycle 32 Day 1: number analyzed (Participants) | 0 | 12
  Cycle 32 Day 1 |  | 0.864 (0.163)
  Cycle 33 Day 1: number analyzed (Participants) | 0 | 10
  Cycle 33 Day 1 |  | 0.870 (0.140)
  Cycle 34 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 34 Day 1 |  | 0.838 (0.160)
  Cycle 35 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 35 Day 1 |  | 0.905 (0.128)
  Cycle 36 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 36 Day 1 |  | 0.779 (0.294)
  Cycle 37 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 37 Day 1 |  | 0.854 (0.170)
  Cycle 38 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 38 Day 1 |  | 0.810 (0.269)
  End of Treatment (EOT): number analyzed (Participants) | 0 | 10
  End of Treatment (EOT) |  | 0.698 (0.324)
  End of Study (EOS): number analyzed (Participants) | 0 | 104
  End of Study (EOS) |  | 0.770 (0.247)

9. Secondary Outcome: Change From Baseline in EQ-5D Health Utility Index Score
Description: as for outcome 8
Time Frame: as for outcome 8
Population: PRO-evaluable population was only consisted of the Australia cohort
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort
Number analyzed (Participants) | 0 | 146
Scores on a scale
  Baseline (Cycle 1 Day 1) |  | 0.786 (0.171)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 139
  Cycle 2 Day 1 |  | 0.013 (0.172)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 132
  Cycle 3 Day 1 |  | 0.021 (0.156)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 119
  Cycle 4 Day 1 |  | 0.052 (0.175)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 113
  Cycle 5 Day 1 |  | 0.052 (0.181)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 106
  Cycle 6 Day 1 |  | 0.037 (0.214)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 105
  Cycle 7 Day 1 |  | 0.033 (0.173)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 97
  Cycle 8 Day 1 |  | 0.050 (0.156)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 94
  Cycle 9 Day 1 |  | 0.057 (0.165)
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 94
  Cycle 10 Day 1 |  | 0.049 (0.192)
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 88
  Cycle 11 Day 1 |  | 0.034 (0.225)
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 84
  Cycle 12 Day 1 |  | 0.029 (0.235)
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 79
  Cycle 13 Day 1 |  | 0.058 (0.203)
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 79
  Cycle 14 Day 1 |  | 0.058 (0.188)
  Cycle 15 Day 1: number analyzed (Participants) | 0 | 74
  Cycle 15 Day 1 |  | 0.062 (0.184)
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 16 Day 1 |  | 0.051 (0.182)
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 17 Day 1 |  | 0.059 (0.165)
  Cycle 18 Day 1: number analyzed (Participants) | 0 | 66
  Cycle 18 Day 1 |  | 0.060 (0.181)
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 62
  Cycle 19 Day 1 |  | 0.061 (0.179)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 61
  Cycle 20 Day 1 |  | 0.069 (0.197)
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 57
  Cycle 21 Day 1 |  | 0.082 (0.169)
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 53
  Cycle 22 Day 1 |  | 0.076 (0.081)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 48
  Cycle 23 Day 1 |  | 0.073 (0.193)
  Cycle 24 Day 1: number analyzed (Participants) | 0 | 42
  Cycle 24 Day 1 |  | 0.085 (0.183)
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 36
  Cycle 25 Day 1 |  | 0.083 (0.192)
  Cycle 26 Day 1: number analyzed (Participants) | 0 | 31
  Cycle 26 Day 1 |  | 0.052 (0.140)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 27
  Cycle 27 Day 1 |  | 0.063 (0.129)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 24
  Cycle 28 Day 1 |  | 0.071 (0.153)
  Cycle 29 Day 1: number analyzed (Participants) | 0 | 21
  Cycle 29 Day 1 |  | 0.056 (0.126)
  Cycle 30 Day 1: number analyzed (Participants) | 0 | 18
  Cycle 30 Day 1 |  | 0.055 (0.122)
  Cycle 31 Day 1: number analyzed (Participants) | 0 | 16
  Cycle 31 Day 1 |  | -0.013 (0.243)
  Cycle 32 Day 1: number analyzed (Participants) | 0 | 12
  Cycle 32 Day 1 |  | 0.049 (0.099)
  Cycle 33 Day 1: number analyzed (Participants) | 0 | 10
  Cycle 33 Day 1 |  | 0.060 (0.098)
  Cycle 34 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 34 Day 1 |  | 0.026 (0.123)
  Cycle 35 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 35 Day 1 |  | 0.092 (0.134)
  Cycle 36 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 36 Day 1 |  | -0.036 (0.240)
  Cycle 37 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 37 Day 1 |  | 0.011 (0.107)
  Cycle 38 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 38 Day 1 |  | -0.012 (0.232)
  End of Treatment (EOT): number analyzed (Participants) | 0 | 10
  End of Treatment (EOT) |  | -0.147 (0.239)
  End of Study (EOT): number analyzed (Participants) | 0 | 104
  End of Study (EOT) |  | -0.022 (0.228)

10. Secondary Outcome: EQ-VAS Score
Description: The EuroQol-5D (EQ-5D) (version 3L) consisted of 2 parts. The second part consisted of a visual analogue scale (the EuroQol-visual analogue scale [EQ-VAS]). The respondent's self-rated health was assessed on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state)
Time Frame: as for outcome 8
Population: PRO-evaluable population was only consisted of the Australia cohort
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort
Number analyzed (Participants) | 0 | 146
Scores on a scale
  Cycle 1 Day 1 |  | 76.9 (16.00)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 137
  Cycle 2 Day 1 |  | 77.3 (15.29)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 132
  Cycle 3 Day 1 |  | 77.4 (15.52)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 119
  Cycle 4 Day 1 |  | 80.3 (14.17)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 113
  Cycle 5 Day 1 |  | 80.4 (14.66)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 107
  Cycle 6 Day 1 |  | 79.8 (15.77)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 105
  Cycle 7 Day 1 |  | 79.7 (14.81)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 99
  Cycle 8 Day 1 |  | 80.1 (13.75)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 95
  Cycle 9 Day 1 |  | 80.9 (14.54)
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 94
  Cycle 10 Day 1 |  | 81.2 (14.75)
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 88
  Cycle 11 Day 1 |  | 81.0 (14.60)
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 84
  Cycle 12 Day 1 |  | 81.3 (13.99)
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 81
  Cycle 13 Day 1 |  | 80.4 (14.37)
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 79
  Cycle 14 Day 1 |  | 80.9 (13.72)
  Cycle 15 Day 1: number analyzed (Participants) | 0 | 74
  Cycle 15 Day 1 |  | 82.1 (12.24)
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 16 Day 1 |  | 82.9 (12.93)
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 17 Day 1 |  | 83.1 (12.89)
  Cycle 18 Day 1: number analyzed (Participants) | 0 | 66
  Cycle 18 Day 1 |  | 83.1 (12.31)
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 62
  Cycle 19 Day 1 |  | 83.7 (12.75)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 62
  Cycle 20 Day 1 |  | 84.5 (12.10)
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 57
  Cycle 21 Day 1 |  | 85.3 (12.03)
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 53
  Cycle 22 Day 1 |  | 85.5 (11.77)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 48
  Cycle 23 Day 1 |  | 84.1 (14.30)
  Cycle 24 Day 1: number analyzed (Participants) | 0 | 42
  Cycle 24 Day 1 |  | 85.6 (12.78)
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 36
  Cycle 25 Day 1 |  | 84.9 (12.89)
  Cycle 26 Day 1: number analyzed (Participants) | 0 | 31
  Cycle 26 Day 1 |  | 87.6 (11.08)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 27
  Cycle 27 Day 1 |  | 88.1 (9.88)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 24
  Cycle 28 Day 1 |  | 87.5 (9.32)
  Cycle 29 Day 1: number analyzed (Participants) | 0 | 21
  Cycle 29 Day 1 |  | 88.5 (9.98)
  Cycle 30 Day 1: number analyzed (Participants) | 0 | 18
  Cycle 30 Day 1 |  | 91.5 (6.97)
  Cycle 31 Day 1: number analyzed (Participants) | 0 | 16
  Cycle 31 Day 1 |  | 88.1 (12.26)
  Cycle 32 Day 1: number analyzed (Participants) | 0 | 12
  Cycle 32 Day 1 |  | 91.0 (8.06)
  Cycle 33 Day 1: number analyzed (Participants) | 0 | 10
  Cycle 33 Day 1 |  | 88.6 (10.61)
  Cycle 34 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 34 Day 1 |  | 91.0 (8.06)
  Cycle 35 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 35 Day 1 |  | 90.0 (11)
  Cycle 36 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 36 Day 1 |  | 87.5 (14.84)
  Cycle 37 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 37 Day 1 |  | 91.5 (7.42)
  Cycle 38 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 38 Day 1 |  | 91.5 (0.71)
  End of Treatment (EOT): number analyzed (Participants) | 0 | 10
  End of Treatment (EOT) |  | 73.6 (23.88)
  End of Study (EOS): number analyzed (Participants) | 0 | 105
  End of Study (EOS) |  | 77.3 (18.99)

11. Secondary Outcome: Change From Baseline in EQ-VAS Score
Description: as for outcome 10
Time Frame: as for outcome 8
Population: PRO-evaluable population was only consisted of the Australia cohort
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort
Number analyzed (Participants) | 0 | 146
Scores on a scale
  Baseline (Cycle 1 Day 1) |  | 76.9 (16.00)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 137
  Cycle 2 Day 1 |  | 0.4 (13.28)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 132
  Cycle 3 Day 1 |  | 0.3 (13.47)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 119
  Cycle 4 Day 1 |  | 2.9 (13.06)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 113
  Cycle 5 Day 1 |  | 3.2 (14.70)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 107
  Cycle 6 Day 1 |  | 2.3 (15.53)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 105
  Cycle 7 Day 1 |  | 2.0 (15.79)
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 99
  Cycle 8 Day 1 |  | 2.4 (13.64)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 95
  Cycle 9 Day 1 |  | 2.3 (12.54)
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 94
  Cycle 10 Day 1 |  | 2.4 (14.44)
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 88
  Cycle 11 Day 1 |  | 2.1 (13.72)
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 84
  Cycle 12 Day 1 |  | 2.9 (13.76)
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 81
  Cycle 13 Day 1 |  | 2.1 (13.84)
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 79
  Cycle 14 Day 1 |  | 2.3 (14.00)
  Cycle 15 Day 1: number analyzed (Participants) | 0 | 74
  Cycle 15 Day 1 |  | 3.5 (12.12)
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 16 Day 1 |  | 3.7 (13.82)
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 70
  Cycle 17 Day 1 |  | 3.9 (12.77)
  Cycle 18 Day 1: number analyzed (Participants) | 0 | 66
  Cycle 18 Day 1 |  | 4.5 (11.86)
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 62
  Cycle 19 Day 1 |  | 4.6 (11.69)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 62
  Cycle 20 Day 1 |  | 5.5 (12.58)
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 57
  Cycle 21 Day 1 |  | 6.0 (11.77)
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 53
  Cycle 22 Day 1 |  | 5.0 (9.71)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 48
  Cycle 23 Day 1 |  | 4.4 (13.20)
  Cycle 24 Day 1: number analyzed (Participants) | 0 | 42
  Cycle 24 Day 1 |  | 4.6 (11.93)
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 36
  Cycle 25 Day 1 |  | 4.3 (10.71)
  Cycle 26 Day 1: number analyzed (Participants) | 0 | 31
  Cycle 26 Day 1 |  | 4.4 (8.63)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 27
  Cycle 27 Day 1 |  | 5.6 (6.26)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 24
  Cycle 28 Day 1 |  | 5.5 (8.24)
  Cycle 29 Day 1: number analyzed (Participants) | 0 | 21
  Cycle 29 Day 1 |  | 5.9 (7.57)
  Cycle 30 Day 1: number analyzed (Participants) | 0 | 18
  Cycle 30 Day 1 |  | 6.5 (7.88)
  Cycle 31 Day 1: number analyzed (Participants) | 0 | 16
  Cycle 31 Day 1 |  | 4.3 (11.52)
  Cycle 32 Day 1: number analyzed (Participants) | 0 | 12
  Cycle 32 Day 1 |  | 7.3 (10.59)
  Cycle 33 Day 1: number analyzed (Participants) | 0 | 10
  Cycle 33 Day 1 |  | 7.1 (12.75)
  Cycle 34 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 34 Day 1 |  | 7.6 (6.68)
  Cycle 35 Day 1: number analyzed (Participants) | 0 | 7
  Cycle 35 Day 1 |  | 6.6 (9.27)
  Cycle 36 Day 1: number analyzed (Participants) | 0 | 6
  Cycle 36 Day 1 |  | 3.5 (8.22)
  Cycle 37 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 37 Day 1 |  | 10.3 (1.71)
  Cycle 38 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 38 Day 1 |  | 9.0 (4.24)
  End of Treatment (EOT): number analyzed (Participants) | 0 | 10
  End of Treatment (EOT) |  | -3.2 (22.24)
  End of Study (EOS): number analyzed (Participants) | 0 | 105
  End of Study (EOS) |  | 0.4 (19.72)

ADVERSE EVENTS:
Time Frame: AEs (serious and non-serious) were recorded on the CRF from the time the participant had taken at least 1 dose of investigational product through and including 28 calendar days after the last administration of the study treatment, an average of 14 months
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Palbociclib+Letrozole India Cohort | Palbociclib+Letrozole Australia Cohort
All-Cause Mortality (participants affected / at risk) | 3/100 | 7/152
Serious Adverse Events (participants affected / at risk) | 18/100 | 45/152
Other Adverse Events (participants affected / at risk) | 85/100 | 151/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib+Letrozole India Cohort (N=100) | Palbociclib+Letrozole Australia Cohort (N=152)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Disease progression (General disorders) | 2 (2) | 6 (6)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2) | 3 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (3)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib+Letrozole India Cohort (N=100) | Palbociclib+Letrozole Australia Cohort (N=152)
Anaemia (Blood and lymphatic system disorders) | 22 (58) | 10 (14)
Neutropenia (Blood and lymphatic system disorders) | 57 (218) | 110 (656)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (34) | 15 (38)
Vision blurred (Eye disorders) | 2 (7) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 10 (12)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 9 (11)
Constipation (Gastrointestinal disorders) | 7 (8) | 32 (45)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 51 (76)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 13 (13)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 34 (50)
Nausea (Gastrointestinal disorders) | 3 (3) | 57 (80)
Vomiting (Gastrointestinal disorders) | 8 (8) | 34 (47)
Asthenia (General disorders) | 8 (9) | 0 (0)
Chest pain (General disorders) | 2 (2) | 13 (19)
Fatigue (General disorders) | 9 (24) | 99 (132)
Influenza like illness (General disorders) | 0 (0) | 14 (17)
Mucosal inflammation (General disorders) | 2 (4) | 33 (61)
Oedema peripheral (General disorders) | 0 (0) | 9 (10)
Pain (General disorders) | 6 (6) | 6 (6)
Pyrexia (General disorders) | 14 (16) | 5 (5)
Gastroenteritis (Infections and infestations) | 0 (0) | 11 (12)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 9 (11)
Nasopharyngitis (Infections and infestations) | 3 (6) | 12 (13)
Oral herpes (Infections and infestations) | 1 (3) | 12 (15)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 57 (87)
Urinary tract infection (Infections and infestations) | 4 (7) | 14 (17)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 10 (11)
White blood cell count decreased (Investigations) | 0 (0) | 15 (23)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 19 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 52 (82)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 35 (49)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 16 (19)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 19 (25)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 23 (32)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 12 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 25 (26)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8)
Dizziness (Nervous system disorders) | 3 (3) | 19 (21)
Headache (Nervous system disorders) | 4 (5) | 47 (71)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 9 (9)
Paraesthesia (Nervous system disorders) | 0 (0) | 11 (12)
Anxiety (Psychiatric disorders) | 0 (0) | 8 (10)
Depression (Psychiatric disorders) | 0 (0) | 8 (8)
Insomina (Psychiatric disorders) | 0 (0) | 18 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 23 (28)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 20 (28)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 14 (21)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (18) | 33 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (12)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 17 (26)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 21 (40)
Hot flush (Vascular disorders) | 0 (0) | 35 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT02679755/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT02679755/SAP_001.pdf